CLINICAL TRIAL: NCT06267092
Title: An Investigation of the Effect of Cagrilintide and Semaglutide Combination Treatment (CagriSema) on Appetite and Functional Brain Activity in People With Overweight or Obesity
Brief Title: A Study of How CagriSema Works on Appetite in People With Excess Body Weight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4944
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A (Other): Participants will not get any medicine during this study.
  Interventions: Other: No treatment given
- Part B (Experimental): Participants will receive CagriSema or placebo (Dose 1,2,3,4) for 16-weeks dose-escalation period followed by 37-weeks intervention period on CagriSema or placebo (Dose 5) that includes a 12-day standardised energy intake period.
  Interventions: Drug: Cagrilintide and Semaglutide; Drug: Placebo

INTERVENTIONS:
Other: No treatment given — Participants will not get any medicine during this study.
  Arms: Part A
Drug: Cagrilintide and Semaglutide — Participants will receive subcutaneous (s.c.) injections of Cagrilintide and Semaglutide.
  Arms: Part B
Drug: Placebo — Participants will receive subcutaneous (s.c.) injections of placebo matched to Cagrilintide and Semaglutide.
  Arms: Part B

SUMMARY:
Part A: The study will look at participants appetite and energy intake and also look at the mechanisms of brain associated with appetite and food intake. Participants will not get any medicine and will be in a group that will be compared to another group receiving a weight-loss medicine. The study will last for about 6 months.

Part B: The study will look at how CagriSema works on participants appetite and energy intake and will be compared with a ''dummy'' medicine. The study will also look at how participants brain works when participants take the medicine. Participants will either get CagriSema or ''dummy'' medicine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-65 years (both inclusive) at the time of signing informed consent
* Right-handed as evaluated by the Edinburgh Handedness Inventory
* Body weight less than or equal to 180 kilogram at screening

For Part A:

* A score of 7 or less on the 16-item Disinhibition subscale of the Three Factor Eating Questionnaire
* Body mass index between 18.5 and 24.9 kilogram per meter square (both inclusive) at screening

For Part B:

* A score of 8 or more on the 16-item Disinhibition subscale of the Three Factor Eating Questionnaire
* Body mass index equal to or above 27.0 kilogram per meter square. Overweight should be due to excess adipose tissue, as judged by the investigator

Exclusion Criteria:

* Contraindication for magnetic resonance scanning

For Part B:

* Glycated haemoglobin greater than or equal to 6.5 % (48 millimoles per mole) at screening
* History of type 1 or type 2 diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Change in mean postprandial appetite score based on visual analogue scale (VAS) | Baseline to week 24
  Measured in millimeter. VAS appetite questions record the participants' sensations within Hunger, Satiety, Fullness and Prospective food consumption by the participants on a paper printed scale line from 0 to 100 mm. The appetite score will be calculated as [hunger + (100 - satiety) + (100 - fullness) + prospective food consumption]/4. Scores of 0 mm are worst and scores of 100 mm are best.

SECONDARY OUTCOMES:
Change in mean postprandial VAS ratings of: hunger, fullness, satiety and prospective food consumption | Baseline to week 24
  Measured in millimeter
Change in average DAILY EATS questionnaire scores over one week for: average hunger, worst hunger, appetite, cravings, satiety and eating drivers index composite score | Baseline pre-treatment ((Day 4 - Day 10) to treatment (Day 156 - Day 162))
  Measured in score points. The DAILY EATS is a 5-item, self-reported measure assessing key eating-related factors (Worst and Average Hunger, Appetite, Cravings, and Satiety). Additionally, an eating drivers index (EDI), comprising the related items Worst Hunger, Appetite, and Cravings can be calculated using this questionnaire. An 11-point numerical rating scale (0-10) is used for each item, with a higher value indicating more hunger, bigger appetite, stronger cravings, or greater satiety.
Change in control of eating questionnaire (COEQ), 4 domains: craving control score, positive mood score, craving for sweets score and craving for savoury food score | Baseline to week 24
  Measured in score points. The COEQ is a self-reported measure assessing various aspects of eating behaviour and related psychological factors. The COEQ has 19 different questions designed to assess the intensity and type of food cravings, as well as subjective sensations of appetite and mood. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control (0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); Higher score represents a greater level of Craving Control.
Change in power of food questionnaire for: food available score, food present score, food tasted score and composite score | Baseline to week 24
  Measured in score points. The power of food questionnaire measures three factors that correspond to different levels of food proximity and reflect responsiveness to food-abundant environments: food available (food that is available, but not physically present), food present (food that is present, but not tasted), and food tasted (food that is tasted, but not consumed). Moreover, an aggregate score is calculated as the mean of the three subdomains. The questionnaire consists of 15 questions, and the participants will be asked to rate their agreement or disagreement with each statement on a 5-point scale (ranging from "strongly disagree" to "strongly agree").
Change in blood oxygen level dependant (BOLD) response to food cues in the brain reward areas | Baseline to week 24
  Measured in percentage
Relative change in total energy intake during ad libitum lunch, evening meal and snackbox | Baseline to week 24
  Measured in percentage
Change in percent energy intake of high fat, sweet food in total ad libitum energy intake in the evening snack box | Baseline to week 24
  Measured in percentage point
Change in total energy intake during ad libitum lunch, evening meal and snackbox | Baseline to week 24
  Measured in kilojoules
Change in total amount of food consumed during ad libitum lunch, evening meal and snackbox | Baseline to week 24
  Measured in grams
Change in body weight | Baseline to week 24
  Measured in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Office dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Charité - Campus Charité Mitte - Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com